CLINICAL TRIAL: NCT01932281
Title: SierraSil as an Ergogenic Aid to Performance in Athletes
Brief Title: SierraSil Joint Formula 14 as an Ergogenic Aid to Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H13-00121
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Muscle Power; Muscle Fatigue
Keywords: muscle power; muscle fatigue; SierraSil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SierraSil (Experimental): SierraSil will be given in a dosage of 3 to 5, 667 mg capsules, according to body weight, daily for 3 weeks.
  Interventions: Dietary Supplement: SierraSil
- Placebo (Placebo Comparator): This is a sugar pill and will be given in a dosage of 3 to 5 capsules daily for 3 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SierraSil — SierraSil is a natural, mineral supplement currently used to improve joint health and function.
  Arms: SierraSil
Dietary Supplement: Placebo — Sugar pill manufactured to mimic SierraSil 667 mg capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether supplementation with SierraSil can improve anaerobic power and reduce muscle fatigue in a group of well-trained athletes.

A secondary purpose is to examine the effect of SierraSil on the severity of delayed onset muscle soreness.

DETAILED DESCRIPTION:
This is a double blind, crossover, pilot study that will examine the effect of SierraSil supplementation on the determinants of human performance. Anaerobic capacity, muscle fatigue, the severity of delayed onset muscle soreness (DOMS) and markers of inflammation will be measured before and after 3 weeks of supplementation with SierraSil or placebo. There will be a 3 week washout period prior to the crossover to ensure SierraSil supplementation has no residual effect.

ELIGIBILITY:
Inclusion Criteria:

* no contraindications to strenuous exercise

Exclusion Criteria:

* muscle or joint injury
* taking any form of anti-inflammatory or pain medication
* females due to the variability that might be introduced due to the phases of the menstrual cycle

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change in total anaerobic capacity | change from baseline at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald C. McKenzie, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada